CLINICAL TRIAL: NCT03158974
Title: A Phase 2, Open-label, Safety, Tolerability, and Efficacy Trial of a Botanical Drug at One Dose Level for the Treatment of External Condylomata Acuminata (Genital Warts) in Adult Immunocompetent Subjects
Brief Title: A Trial of a Botanical Drug Containing East Indian Sandalwood Oil (EISO) for the Treatment of External Genital Warts
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated study due to financial constraints.
Sponsor: ViroXis Corporation (Industry)
Collaborators: Progressive Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIR007-01
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Condylomata Acuminata
Keywords: External Genital Warts
MeSH Terms: conditions — Condylomata Acuminata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VIR007 (Experimental): Cream containing 10% East Indian Sandalwood Oil (EISO)/Albuterpenoids
  Interventions: Drug: East Indian Sandalwood Oil Cream

INTERVENTIONS:
Drug: East Indian Sandalwood Oil Cream — Cream containing 10% East Indian Sandalwood Oil (EISO)/Albuterpenoids
  Other Names: VIR007

SUMMARY:
This trial will be a phase 2, open-label, study to evaluate the safety, tolerability, and efficacy of VIR007 when administered topically for up to 60 days to adults between the ages of 18 to 65 years with a clinical diagnosis of external condylomata acuminata.

DETAILED DESCRIPTION:
This trial will be a phase 2, open-label, study to evaluate the safety, tolerability, and efficacy of VIR007 when administered topically for up to 60 days to adults between the ages of 18 to 65 years with a clinical diagnosis of external condylomata acuminata.

Subjects will enter the Screening Period once the informed consent process has been completed. Subjects with a clinical diagnosis of external condylomata acuminata and who meet all inclusion and none of the exclusion criteria will be enrolled.

Once subject eligibility is confirmed and the screening procedures completed, the subject will start the Treatment Period of the study. All enrolled subjects will receive VIR007 (cream containing 10% EISO) with the first dose applied topically during Visit 1 (Day 1). Subjects will be instructed on how to apply the study medication twice daily for up to 60 days or until the Investigator determines the lesions have cleared. Subjects will return to the clinic for study-related assessments on Study Days 7, 14, 28, 42 and a Final Study Visit on Day 60. 30 days following complete resolution, as determined by the study investigator, or, on Study Day 90, subjects will receive a follow-up telephone call and be queried regarding condition status since study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Are ≥18 but ≤65 years of age
2. Are in good general health, as confirmed by medical history
3. Have a clinical diagnosis of condylomata acuminata with ≥2 but ≤10 visible external genital warts (EGWs)
4. Have EGW lesions <200mm2
5. Are free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of adverse events.
6. Must be willing to use a barrier method of birth control while enrolled in the study.
7. If female of childbearing potential, must have a negative urine pregnancy test result prior to study treatment and must be willing to use a barrier method of birth control while enrolled in the study.
8. Are willing to refrain from using any lotions, moisturizer, cleansers, cosmetics or creams, other than those issued as part of the study, on the affected areas during the treatment period.
9. Are able to give written informed consent in a manner approved by the Institutional Review Board or Ethics Review Committee and comply with the requirements of the study.
10. Are willing to avoid participation in any other clinical trial for the duration of this study.
11. Are willing and able to participate as an outpatient, making regularly scheduled visits to the study center during the treatment and to comply with all study requirements including concomitant medication and other treatment restrictions.
12. Are willing to forgo all other treatments (prescription, nonprescription, and nutritional supplements) for their EGWs.

Exclusion Criteria:

1. Have evidence of an active malignancy or have been immunocompromised within the 60 days prior to Screening.
2. Received any treatment for their EGW within 60 days of planned study enrollment.
3. Are pregnant, breast-feeding, or planning to become pregnant during the study.
4. Have EGWs ≥200mm2.
5. Have any evidence, currently or in the last 60 days, of herpes genitalis or any other current and/or recurrent genital or uncontrolled infection that, in the opinion of the investigator, could confound the results of the study including human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C.
6. Have any abnormal skin conditions, body piercings, hypertrophic scarring or body modification in the area that, in the opinion of the investigator, might affect the accurate evaluation of EGWs.
7. Shares a household with a subject currently enrolled in the study.
8. Have any condition that, in the opinion of the investigator, would confound the safety and/or efficacy assessments.
9. Have internal genital wart lesions, including the urethra, vagina and/or rectum.
10. If female, have any evidence of cervical dysplasia.
11. Have evidence of clinically significant or unstable disease (eg, stroke, heart attack).
12. Have a known sensitivity to any of the constituents of the test product including sensitivities to sandalwood oil, fragrances or any member of the Compositae family of vascular plants (eg, sunflowers, daisies, dahlias, etc.).
13. Have a history of Bowenoid papulosis.
14. Have received any of the following within 90 days prior to study treatment:

    * Interferon or interferon inducers
    * Cytotoxic drugs
    * Immunomodulators or immunosuppressive therapies (inhaled/intranasal corticosteroids are permitted)
    * Oral or parenteral corticosteroids
    * Topical corticosteroids if greater than 2 gm/day
    * Any dermatologic procedures or surgeries on the study area (including EGW treatments)
15. Have a history of alcohol abuse, or suspected alcohol abuse, in the past two years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-17 (Actual); Study Completion 2018-06-17 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 60-days
  Safety will be assessed by evaluating adverse events (AEs) with respect to severity, duration, and relationship to study drug.

SECONDARY OUTCOMES:
Incidence of treatment-emergent tolerability issues | 60-Days
  Tolerability will be assessed by the number of subjects reporting discomfort either during or immediately following the application of VIR007
Percentage of patients achieving complete clearance | 60-days
  The percentage of subjects achieving complete clearance of all EGW lesions over the course of the trial
Time to clearance | 60-days
  Time to clearance over the trial
Remission | 90-days
  Percentage of subjects continuing in remission at the follow-up call

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lee, MD, Principal Investigator — Progressive Clinical Trials
Locations (1):
- Progressive Clinical Research, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No